CLINICAL TRIAL: NCT04106102
Title: Study of the Effectiveness of Transcranial Direct Current Stimulation on Obsessive Compulsive Disorder
Acronym: EFFI-STOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-API-02
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcramial Direct current stimulation (Active Comparator): Implement of Transcramial Direct current stimulation
  Interventions: Device: Transcramial Direct current stimulation
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Transcramial Direct current stimulation — Two sessions of 5 stimulations will be made on patient with obsessive-compulsive disorder
  Arms: Transcramial Direct current stimulation
Device: Placebo — Two sessions of 5 stimulations will be made on patient with obsessive-compulsive disorder without direct current. They xwill just wear electrodes.
  Arms: Placebo

SUMMARY:
The usual management of Obsessive Compulsive Disorders is based on cognitive-behavioural psychotherapy, as well as the use of serotonergic antidepressants. Nevertheless, a significant proportion of patients (40% to 60%) are non-responders to these conventional therapies, and remain severely handicapped.

transcranial Direct current stimulation (tDCS) has already proven its effectiveness, in addition to drug approaches, in various clinical settings, such as depression or acoustic-verbal hallucinations. This technic appears to be an extremely interesting alternative This is a non-invasive neuromodulation technique (application of a low intensity direct current (1 to 2 mA) between two electrodes positioned on the scalp) that allows the neural activity of different brain areas to be modulated simultaneously. It is a simple and inexpensive technique with excellent tolerance.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a common psychiatric condition (prevalence 2-3%), with a chronic course, and significantly impairs the quality of life and functioning of sufferers quality of life and functioning. Cognitive-behavioral psychotherapies are the standard treatment, and the use of serotonergic antidepressants. Nevertheless, a significant proportion of patients (40% to 60%) are non-responders to these conventional therapies, and remain severely handicapped (Pallanti & Quercioli, 2006).

Recent advances in neuroimaging techniques have enabled us to pinpoint the neuroanatomical basis of OCD. of OCD, notably involving dysfunctions affecting cortico-striato-pallido-thalamocortical circuits.

This knowledge of the pathophysiology of the disease has led to the development of focal intervention strategies, aimed at modulating the activity of these cortico-subcortical loops in order to reduce obsessive-compulsive symptomatology, using invasive (deep brain stimulation via stereotactic electrode implantation) or non-invasive (repeated trancranial magnetic stimulation or rTMS) procedures or rTMS). In the case of rTMS, recent studies have demonstrated the efficacy of a single treatment in patients with resistant OCD. the efficacy of low-frequency stimulation of the pre-supplementary motor area (pre-SMA), a brain area involved in cognitive inhibition processes. However, these methods have limitations invasive nature in the case of deep brain stimulation, and the need for an expensive technical for rTMS.

There is therefore a clear need to develop new therapeutic approaches for OCD, combining efficacy efficacy, safety and patient acceptance.

In this context, transcranial direct current stimulation (tDCS) is an extremely interesting alternative. This non-invasive neuromodulation technique involves applying a low-intensity direct current current (1 to 2 mA) between two electrodes positioned on the scalp. It enables modulate neuronal activity in different brain areas simultaneously. It also has the advantage of being the advantage of simple, low-cost use, as well as excellent tolerance.

TDCS has already provided evidence of its efficacy, as a complement to medication-based approaches, in a variety of clinical contexts, such as depression (Kalu et al., 2012) or acoustic-verbal hallucinations (Brunelin et al., 2012).

With regard to OCD, preliminary data, in the form of case reports (Narayanaswamy & al., 2015; Mondino & al., 2015) and open studies (Bation & al., 2016), appear very promising. In Bation & al.'s study, in 8 patients with drug-resistant OCD, tDCS led to an average 26.4% reduction in symptoms (measured by the Y-BOCS scale).

There is currently no consensus regarding electrode positioning for the treatment of OCD, but studies suggest (Senço & al., 2015) that a set-up combining the cathode opposite the pre-supplementary motor area motor area and the anode in an extracephalic position (right deltoid) would modulate the brain regions involved in the pathophysiology of OCD.

We propose to study the efficacy and tolerability of tDCS in the treatment of drug-resistant OCD in a in a randomized, controlled, prospective, double-blind trial. To the best of our knowledge, this is the first trial of this type for tDCS in this condition.

ELIGIBILITY:
Inclusion Criteria:

* Presenting an obsessive-compulsive disorder according to the criteria of Diagnostic and Statistical Manual of Mental Disorders 5, evolving for at least two years
* Of significant clinical intensity: Yale-Brown's obsession-compulsion scale ≥ 16/40 continuously over the last 6 months. This criteria of persistent severity over the last 6 months will be explored by an in-depth clinical interview at the inclusion visit (Baseline BL)
* Resistant despite treatment with: 2 serotonergic antidepressants, each received for at least 8 weeks, at the maximum recommended or tolerated dosage AND behavioural and cognitive therapy for at least 6 months
* Drug treatment unchanged for at least 12 weeks

Exclusion Criteria:

* Patient with psychotic disorder, bipolar mood disorder, substance abuse or dependence (excluding tobacco)
* Patient at risk of suicide (score ≥ 2 on item 10 of the Montgomery-Åsberg depression rating scale)
* Contraindications to the practice of transcranial direct stimulation : history of cerebral pathology, intracranial hypertension, neurosurgery, cephalic metal implant, pacemaker
* Unbalanced epilepsy
* Previous use of transcranial direct stimulation (problem of maintaining the integrity of the blind procedure)
* Pregnancy or breastfeeding in progress, woman in a state of procreation without effective contraception (a urine pregnancy test will be performed)
* Scalp skin pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown's obsession-compulsion scale (Y-BOCS) | 3 month
  The evolution (continuous parameter) of this score between the beginning of treatment (Baseline BL) and the visit at 3 month will be calculated.
  The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) is a scale for assessing obsessive symptomatology scale for assessing obsessional symptomatology. It is reliable, accurate and sensitive to therapeutic changes. The French version is well validated. It allows comprehensive assessment and repeated measurement of two types of target symptoms target symptoms: obsessions (score from 0 to 20) and compulsions (score from 0 to 20), leading to an overall severity score of 0 to 40. Developed since 1989, it is the reference measure of OCD in therapeutic studies. A score of 16 or more is frequently used to select obsessive-compulsive subjects for controlled controlled studies.
  This is a hetero-questionnaire administered in the form of a structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno GIORDANA, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France